CLINICAL TRIAL: NCT00807586
Title: SAAB: Randomized, Double Blind STudy of Corticosteroid Pulse After Ablation
Brief Title: Corticosteroid Pulse After Ablation
Acronym: SAAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ep002
Record Dates: First submitted 2008-12-10; First posted 2008-12-12 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Corticosteroid; Radiofrequency catheter ablation for atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Steroid (Experimental)
  Interventions: Drug: Solumedrol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solumedrol — 100mg, given once within 2 hours of the end of the ablation procedure
  Arms: Steroid
Drug: Placebo — Normal saline (1.6 cc)
  Arms: Placebo

SUMMARY:
Radiofrequency ablation is an effective treatment for atrial fibrillation. However, about 20% of the time the atrial fibrillation recurs. Steroids given after the ablation may decrease inflammation caused by the ablation and thus improve healing and decrease the chance of recurrence of atrial fibrillation.

In this study patients will be randomized to receive intravenous steroids or not immediately following the ablation.

DETAILED DESCRIPTION:
Atrial fibrillation, a common arrhythmia, is the source of considerable morbidity. Prevalence of atrial fibrillation in adults is 0.5%, increasing to 10% in those patients over the age of seventy five. Numbers are expected to increase nearly 2.5 fold over the next 50 years. Radiofrequency (RF) ablation to cure atrial fibrillation has become an established and effective therapy in the many atrial fibrillation patients. However, approximately 20% return with recurrent atrial fibrillation after ablation.

RF ablation directly targets the substrate for atrial fibrillation, cauterizing cardiac tissue through the application of radiofrequency energy , causing a myocardial lesion which effectively blocks the errant pathway. This process of RF ablation induces an inflammatory effect. As the lesion heals it often enlarges. This may contribute to recurrence of atrial fibrillation after ablation, as well as increased pain. There is some early evidence that a single dose of corticosteroids after ablation may improve the healing process, thus decreasing pain and incidence of recurrent atrial fibrillation.

The aim of the study is to determine the usefulness of a one time dose of solumedrol following radiofrequency ablation for atrial fibrillation..

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Drug refractory, symptomatic paroxysmal atrial fibrillation

Exclusion Criteria:

* Contraindication to solumedrol
* Persistent or permanent Atrial Fibrillation
* Previous history of radiofrequency ablation for atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Melby, MD, Principal Investigator — Minneapolis Heart Institute
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Grubb NR, Furniss S. Science, medicine, and the future: Radiofrequency ablation for atrial fibrillation. BMJ. 2001 Mar 31;322(7289):777-80. doi: 10.1136/bmj.322.7289.777. No abstract available. PMID 11282867
- [Background] Pappone C, Santinelli V. Atrial fibrillation ablation: state of the art. Am J Cardiol. 2005 Dec 19;96(12A):59L-64L. doi: 10.1016/j.amjcard.2005.09.063. Epub 2005 Oct 5. PMID 16399094
- [Background] Fenelon G, Franco M, Mora O, Katchburian E, de Paola AA. Combined therapy with steroids and antioxidants prevents ultrastructural damage surrounding chronic radiofrequency lesions. Pacing Clin Electrophysiol. 2004 Jan;27(1):65-72. doi: 10.1111/j.1540-8159.2004.00387.x. PMID 14720157
- [Background] Fenelon G, Fernandes R, Franco M, de Paola AA. Steroids prevent late extension of radiofrequency lesions in the thigh muscle of infant rats: implications for pediatric ablation. J Interv Card Electrophysiol. 2003 Aug;9(1):7-13. doi: 10.1023/a:1025308218103. PMID 12975564

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Steroid | Placebo
Started | 60 | 59
Completed | 54 | 58
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid | Placebo | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (10.2) | 60.0 (11.4) | 60.1 (11.2)
Sex/Gender, Customized [Number; unit: participants]
  Female | 14 | 13 | 27
  Male | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Atrial Arrhythmias at 6 Weeks
Description: Clinically significant atrial arrhythmias include ER, urgent care, or hospitalization for atrial fibrillation, cardioversion for atrial fibrillation, or atrial fibrillation requiring an increase in anti-arrhythmia medication
Time Frame: 6 weeks
Population: 3 patients lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 58 | 58
Participants | 4 | 12

2. Secondary Outcome: Cardiac Pain Assessment
Description: Perception of cardiac pain assessed by a numerical pain scale (0= no pain; 10=worst pain imaginable)
Time Frame: one day and one week
Population: 4 patients lost to follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 58 | 57
units on a scale
  Pain Scale Day 1 | 0.9 (1.5) | 1.5 (2.4)
  Pain Scale Week 1 | 0.8 (1.9) | 0.6 (1.2)

3. Secondary Outcome: Symptoms Post Ablation Requiring Diuretic
Description: Occurrence of shortness of breath or edema requiring administration of a diuretic
Time Frame: 6 weeks
Population: Data were not collected on this outcome
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Repeat Intervention
Description: Need for repeat ablation
Time Frame: 3 months
Population: 14 patients lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Steroid | Placebo
Number analyzed (Participants) | 50 | 55
Participants | 2 | 8

ADVERSE EVENTS:
Time Frame: there were Adverse Events collected from six weeks to 1 year
Arm/Group | Steroid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/59
Other Adverse Events (participants affected / at risk) | 25/60 | 17/59
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid (N=60) | Placebo (N=59)
Atrial Flutter (Cardiac disorders) | 5 (5) | 3 (3)
Chest Pain (Cardiac disorders) | 1 (1) | 5 (5)
Shortness of Breath (Cardiac disorders) | 7 (7) | 2 (2)
Fatigue (Cardiac disorders) | 6 (6) | 1 (1)
Back Pain (Cardiac disorders) | 3 (3) | 0 (0)
Edema/fluid overload (Cardiac disorders) | 3 (3) | 1 (1)
Hypotension (Cardiac disorders) | 0 (0) | 3 (3)
Abdominal Pain (Cardiac disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
This was a single center study trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No